CLINICAL TRIAL: NCT07187063
Title: Using Urine Tumor DNA to De-Intensify Surveillance in Non-Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20233622
Record Dates: First submitted 2025-08-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- De-Intensified Arm (Experimental): Less-frequent cystoscopy surveillance
  Interventions: Diagnostic Test: UroAmp Test (Convergent Genomics, Inc.)
- Standard Surveillance Arm (No Intervention): Regular follow-ups and standard care

INTERVENTIONS:
Diagnostic Test: UroAmp Test (Convergent Genomics, Inc.) — Non-invasive genomic urine test that can reliably detect, monitor, and predict the risk of urothelial cancer or its recurrence, potentially before signs and symptoms develop or become detectable by historical standards of care.
  Arms: De-Intensified Arm

SUMMARY:
The goal of this clinical trial is to use urine tumor DNA (utDNA) as an indicator for non-muscle invasive bladder cancer to identify patients suitable for less frequent cystoscopy surveillance.

ELIGIBILITY:
Inclusion Criteria:

* AUA high-risk bladder cancer1
* Received induction BCG or gemcitabine/docetaxel
* Negative initial post-induction therapy assessment (negative cytology and cystoscopy +/- biopsy)

Exclusion Criteria:

* High-risk NMIBC within 3 years
* Prior induction intravesical therapy
* Variant histology
* Concurrent upper tract disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of cystoscopies | From enrollment to 24 months
  The rate of cystoscopies (cystoscopies per month), compared between the De-intensified and the standard surveillance arms, is the primary outcome measure.

SECONDARY OUTCOMES:
Event-free survival | From enrollment to 24 months
  An event is defined as: high-grade recurrence, progression to muscle invasive disease, or metastatic disease
Recurrence-free survival | From enrollment to 24 months
  We will compare the rate of any recurrences (including low-grade) between the De-intensified and the standard surveillance groups
Patient-reported outcomes | From enrollment to 24 months
  The National Comprehensive Cancer Network Distress thermometer and the European Organisation For Research And Treatment Of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Non-Muscle Invasive Bladder Cancer (NMIBC-24) Module will be collected and compared between study arms

OTHER OUTCOMES:
Interim Analysis | 3 months
  After 50% enrollment, the rate of conversion from low-risk on the utDNA test to high risk will be evaluated at 3 months. If this rate exceeds 50%, the study will be terminated for futility.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Clements, MD, MS, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Considering whether to involve other sites in the trial

REFERENCES:
- [Background] Clinical Trials in Progress: Bladder Cancer: Monday, April 28, 9-11 am. Journal of Urology. https://doi.org/10.1097/01.JU.0001110440.53375.7d
- [Background] Salari K, Sundi D, Lee JJ, Wu S, Wu CL, DiFiore G, Yan QR, Pienkny A, Lee CK, Oberlin D, Barme G, Piser J, Kahn R, Collins E, Phillips KG, Caruso VM, Goudarzi M, Garcia-Ransom M, Lentz PS, Evans-Holm ME, MacBride AR, Fischer DS, Haddadzadeh IJ, Mazzarella BC, Gray JW, Koppie TM, Bicocca VT, Levin TG, Lotan Y, Feldman AS. Development and Multicenter Case-Control Validation of Urinary Comprehensive Genomic Profiling for Urothelial Carcinoma Diagnosis, Surveillance, and Risk-Prediction. Clin Cancer Res. 2023 Sep 15;29(18):3668-3680. doi: 10.1158/1078-0432.CCR-23-0570. PMID 37439796
- [Background] Bicocca VT, Phillips KG, Fischer DS, Caruso VM, Goudarzi M, Garcia-Ransom M, Lentz PS, MacBride AR, Jensen BW, Mazzarella BC, Koppie T, Korkola JE, Gray JW, Levin TG. Urinary Comprehensive Genomic Profiling Correlates Urothelial Carcinoma Mutations with Clinical Risk and Efficacy of Intervention. J Clin Med. 2022 Sep 30;11(19):5827. doi: 10.3390/jcm11195827. PMID 36233691
- See also: Patient-oriented presentation on the study — https://sites.google.com/view/deintensifyutdna/home?authuser=0